CLINICAL TRIAL: NCT06712680
Title: A Phase I/II , Open-label, Multi-center, Multi-cohort Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of HYP-6589 Monotherapy in Advanced Solid Tumors and Combination With Tyrosine Kinase Inhibitors in Patients With Advanced NSCLC With Target-driven Gene Positivity
Brief Title: A Phase I/II Study of HYP-6589 Monotherapy in Treating Advanced Solid Tumors and in Combination With Tyrosine Kinase Inhibitors in Treating Patients With Advanced NSCLC Positive for Driver Genes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY0006-101
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product HYP-6589 (Experimental): HYP-6589 should be administered orally at the recommended dosage
  Interventions: Drug: Test Product HYP-6589

INTERVENTIONS:
Drug: Test Product HYP-6589 — HYP-6589 should be administered orally at the recommended dosage

SUMMARY:
This is a multi-center , open-label, phase 1/2 study to evaluate the safety, efficacy, and pharmacokinetic (PK) characteristics of HYP-6589 in monotherapy in advanced solid tumors and combination with tyrosine kinase inhibitors in patients with advanced NSCLC with target-driven gene positivity.

DETAILED DESCRIPTION:
The study starts with a dose escalation part (Part 1) followed by a dose expansion part (Part 2). The main purpose of this study is to evaluate the safety and tolerability of the drug HYP-6589 and determine the maximum tolerated dose (MTD) (if any) and/or the recommended dose(s) (RD) and preliminary anti-tumor activity. Additional purposes of the study are to evaluate the pharmacokinetics (PK) properties.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign an informed consent form, understand the study and be willing and able to follow and complete all trial procedures;
* ≥18 years old and ≤80 years old, gender: male or female;
* Histological or cytological confirmation of unresectable and/or metastatic advanced solid tumors;
* At least one measurable lesion (according to RECIST 1.1 version);
* Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
* Life expectancy ≥3 months;
* Participant must have adequate main organ function;
* Fertile female patients must have a negative serological pregnancy test within 7 days before the first dosing and be willing to use effective birth control/contraception to prevent pregnancy during the study period up to 6 months after the last dosing of the study. Male patients must agree to have no sperm donation plans and to use effective contraceptive methods during the study period until 6 months after the last dose of the study. Postmenopausal women must have amenorrhea for at least 12 months before they are considered infertile.

Exclusion Criteria:

* Participants who have received other investigational drugs or participated in interventional medical device studies within 4 weeks prior to the first administration of the study drug;
* Participants who have received (attenuated) live vaccines within 4 weeks prior to the first administration of the study drug;
* Participants who have undergone major organ surgery (excluding biopsy) within 4 weeks prior to the first administration of the study drug or have experienced significant trauma, or who require elective major organ surgery (excluding biopsy) during the study period;
* Participants who, based on computerized tomography (CT) or magnetic resonance imaging (MRI) examinations conducted during the screening period and before radiological assessment, have uncontrolled, unstable, or active central nervous system (CNS) metastases;
* Participants with clinically uncontrollable hypertension (defined in this protocol as having a systolic blood pressure > 150 mmHg and/or a diastolic blood pressure > 100 mmHg despite antihypertensive treatment, and which is considered clinically significant by the investigator);
* Participants who have received allogenic tissue/organ transplants in the past;
* Participants with active infections deemed inappropriate for entry into the study by the investigator;
* Participants with uncontrolled third-space effusion requiring clinical intervention;
* Participants with a history of drug abuse or medical, psychological, or social conditions that may interfere with study participation or impair the assessment of study outcomes;
* Participants with known gastrointestinal (GI) dysfunction or GI diseases that are likely to significantly affect the absorption or metabolism of oral medications (e.g., dysphagia, active upper gastrointestinal ulcer, intestinal obstruction, nausea, vomiting, and diarrhea of grade 3 or higher that persist despite optimal supportive care within 3 days);
* Participant whose toxicities from previous anti-cancer therapy have not resolved, defined as toxicity (hair loss excluded) that has not resolved to grade ≤1 (CTCAE 5.0 version, peripheral neuropathy, ≤grade 2; exclusion criteria specified);
* Female participants who are breastfeeding or have positive urine or blood pregnancy test results during the screening period; female participants who have a planned pregnancy, sperm donation, or egg donation during the study period or within 6 months after the last study drug administration;
* Known history of hypersensitivity to any of the components of the test formulation.
* Participants who have had other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma of the skin;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2028-04-10 (Estimated); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation (Part One): Incidence and Nature of Dose-Limiting Toxicity (DLT) | 24 days during the first 4-week cycle
  Dose-Limiting Toxicity (DLT) will be defined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose Escalation (Part One): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Dose Escalation (Part One): Other safety indicators | Up to 2 years
  Adverse events (AE), physical examination, vital signs, electrocardiogram (ECG) and laboratory test results that occur during the treatment
Dose Expansion (Part Two): Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants who have a confirmed Complete Response (CR) or a Partial Response (PR)

SECONDARY OUTCOMES:
Dose Expansion (Part Two): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | Up to 2 years
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Dose Expansion (Part Two): Other safety indicators | Up to 2 years
  Adverse events (AE), physical examination, vital signs, electrocardiogram (ECG) and laboratory test results that occur during the treatment.
Dose Escalation and Expansion: Assessment of HYP-6589 Cmax | Up to 2 years
  Maximum concentration observed (Cmax) observed from the pharmacokinetic profile
Dose Escalation and Expansion: Assessment of HYP-6589 AUC | Up to 2 years
  Area under the concentration versus time curve calculated using the trapezoidal method
Dose Escalation and Expansion: Assessment of HYP-6589 T1/2 | Up to 2 years
  The time it takes for half the drug concentration to be eliminated calculated using slope of the terminal line
Dose Escalation (Part One): Objective Response Rate (ORR) | Up to 2 years
  Proportion of participants who have a confirmed complete response (CR) or a Partial Response (PR) determined by Investigator per the Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1
Dose Escalation and Expansion: Duration Of Response (DOR) assessed by investigator per Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 | Up to 2 years
  Duration Of Response (DOR) is defined as the time from the measurement criteria are first met for complete response (CR) /Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease.
Dose Escalation and Expansion: Disease Control Rate (DCR) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Disease Control Rate is defined as the percentage of participants who have achieved CR or PR or have demonstrated stable disease
Dose Escalation and Expansion: Progression-Free Survival (PFS) assessed by investigator per RECIST Version 1.1 | Up to 2 years
  Progression-Free Survival (PFS) is defined as the time from the date of first administration of HYP-6589 to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 or death from any cause, whichever occurs first
Dose Escalation and Expansion: Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) is defined as the time from the date of first administration of HYP-6589 to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China